CLINICAL TRIAL: NCT03331458
Title: Physical Activity in Men Newly Diagnosed With Prostate Cancer: A Feasibility Study
Acronym: PACMen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00083320
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: physical activity
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subjects with prostate cancer (Experimental)
  Interventions: Behavioral: exrecise intervention

INTERVENTIONS:
Behavioral: exrecise intervention — Subjects will undergo pre-intervention measures, complete a daily physical activity diary, and post-intervention measures

SUMMARY:
Recent research has indicated that physical activities incorporating moderate-intensity exercise can be safely performed during treatment and substantially reduces treatment-related side effects, such as fatigue, sleep disturbances, cognitive impairment, and nausea. However, little is known about physical activity levels prior to treatment and whether providing an exercise intervention pre-treatment may improve functional capacity during treatment.

The purpose of this study is to

1. Measure physical activity levels and functional capacity in men newly diagnosed with prostate cancer prior to treatment and
2. Explore whether a 2-week physical activity intervention is feasible during the pre-treatment timeframe:

   1. Examine intervention safety and tolerance by self-report
   2. Examine changes in functional capacity by 6-minute walk test
   3. Examine changes in symptom experience by self-report

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with prostate cancer
* will not start treatment for at least 2 weeks
* able to read and understand English
* capable of giving informed consent
* at least 18 years old

Exclusion Criteria:

* patients who are incompetent for interview (documented diagnosis of active psychosis or dementia)
* unable to provide informed consent as assessed by the interviewer
* too sick to participate, as judged by a member of the research team or the exercise physiologist
* have been treated for another cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute walk test | baseline, 2 weeks post intervention
  Distance walked in 6 minutes
Change in balance test | baseline, 2 weeks post intervention
  Ability to balance
Change in time up to go test | baseline, 2 weeks post intervention
  Time to get up from chair, walk 30 meters and return to sit in chair
Change in Godin Leisure Time Score | baseline, 2 weeks post intervention
  physical activity score
Change in rate of perceived exertion | baseline, 2 weeks post intervention
  physical exertion score
Change in metabolic equivalent | baseline, 2 weeks post intervention
  metabolic activity score
Change in distress score | baseline, 2 weeks post intervention
  distress score
Change in self-efficacy score | baseline, 2 weeks post intervention
  self-efficacy score
Change in symptom inventory score | baseline, 2 weeks post intervention
  description of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Allen, Principal Investigator — Duke University
Locations (1):
- Duke Raleigh Cancer Center, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share feasibility study data